CLINICAL TRIAL: NCT04342741
Title: A Comparison Between Inpatient and Outpatient Balloon Catheter Cervical Ripening: A Prospective Randomized Controlled Trial
Brief Title: Inpatient and Outpatient Balloon Catheter Cervical Ripening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Rahana Abd Rahman, Co-primary investigator, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FF-2017-358
Record Dates: First submitted 2020-04-07; First posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Caesarean Section; Infection
Keywords: cervical ripening; Foley catheter; Patient satisfaction
MeSH Terms: conditions — Infections; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: The patients were randomised to cervical ripening with foley catheter as inpatient or outpatient setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foley catheter inpatient (Active Comparator): Participants had intracervical ripening with foley catheter after admission into the ward.
  Interventions: Device: Foley catheter cervical ripening
- Foley catheter outpatient (Active Comparator): Participants had intracervical ripening with foley catheter and allowed home.
  Interventions: Device: Foley catheter cervical ripening

INTERVENTIONS:
Device: Foley catheter cervical ripening — Participants were assessed when labour was established or the following morning.

SUMMARY:
A randomised controlled trial comparing cervical ripening using foley catheter as in- or outpatient setting.

DETAILED DESCRIPTION:
The study evaluated the efficacy and safety of outpatient versus inpatient Foley catheter cervical ripening and patients' satisfaction. Sixty low-risk women were randomized to outpatient and inpatient management of intracervical Foley catheter digital insertion. The outpatient group was provided with verbal and written 24-hours contact information and instructions. Both groups were reassessed the next morning unless labor had begun or the catheter had dropped off.

ELIGIBILITY:
Inclusion Criteria:

* singleton
* gestational age beyond 37 weeks
* cephalic presentation
* intact membranes
* Bishop score less than 6
* lives within 10km from National University Malaysia Medical Centre or able to reach within 30 minutes
* readily available transport

Exclusion Criteria:

* intrauterine death
* intrauterine fetal growth restriction
* estimated fetal weight more than 4000gram
* fetal anomalies
* abnormal pre-induction cardiotocograph
* non-vertex presentation
* unstable lie
* sepsis
* hypertension
* allergy to latex
* previous uterine scar
* history of antepartum haemorrhage
* parity of 6 and more
* placenta praevia
* suspected cephalopelvic disproportion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Caesarean section rate | From the time of recruitment until delivery
  Percentage of Caesarean section
Neonatal sepsis | From birth up to 30 days
  Percentage of neonates with sepsis

SECONDARY OUTCOMES:
Maternal age | At the time of recruitment
  Mean maternal age in years
Ethnicity | At the time of recruitment
  Percentage of each races
Education level | At the time of recruitment
  Percentage of participants with secondary or higher education level
Occupation | At the time of recruitment
  Percentage of participants who were professional or non professional or housewives
Pre-pregnancy maternal body mass index | At the time of recruitment
  Mean pre-pregnancy body mass index in kg/m2
Parity | At the time of recruitment
  Percentage of participants who are nulliparous or multiparous
Gestation at recruitment | At the time of recruitment
  Percentage of participants who were recruited at 40 or 40 weeks and 10 days
Indication | At the time of recruitment
  Percentage of participants who were induced based on indication
Bishop score pre-induction | Pre-intervention
  Mean Bishop score prior to induction. Unfavourable score has minimum score of 0 and maximum score of 5.
Bishop score at second assessment | From insertion of Foley catheter until labour established or the following morning
  Mean Bishop score at second assessment. Unfavourable score has minimum score of 0 and maximum score of 5.
Management at second assessment | At time of recruitment until delivery
  Percentage of participants who had dinoprostone insertion or artificial rupture of membranes
Duration from induction until favourable Bishop score | At time of recruitment until delivery
  Mean duration taken from induction until favourable Bishop score in hours
Augmentation with oxytocin | At time of recruitment until delivery
  Percentage of participants who required oxytocin augmentation
Duration of oxytocin use | At time of recruitment until delivery
  Mean duration of oxytocin use in minutes
Duration from amniotomy until delivery | At time of recruitment until delivery
  Mean duration from amniotomy until delivery in hours
Duration from induction until delivery | At time of recruitment until delivery
  Mean duration from induction until delivery in hours
Delivery within 24 hours | At time of recruitment until delivery
  Percentage of participants who delivered within 24 hours from induction
Duration of inpatient stay | At time of recruitment until delivery
  Mean duration of inpatient stay in hours
Total blood loss | At the time of delivery
  Median blood loss in millilitres
Intrapartum pyrexia | At the time of delivery
  Percentage of participants with intrapartum pyrexia
Primary postpartum haemorrhage | Immediately at delivery up to 42 days
  Percentage of participants with primary postpartum haemorrhage
Birth weight | At the time of delivery
  Mean birth weight in grams
Arterial cord blood acidity or alkalinity | At the time of delivery
  Mean arterial cord blood acidity or alkalinity
Neonatal white cell count | At the time of delivery
  Mean neonatal white cell count in liter
Neonatal C-reactive protein | At the time of delivery
  Median neonatal C-reactive protein in milligram per liter
Discomfort with foley catheter | At the time of recruitment until active phase of labour
  Percentage of participants experienced discomfort with foley catheter
Ability to cope with discomfort | At the time of recruitment until active phase of labour
  Percentage of participants able to cope with discomfort
Intention to use the method again | Through study completion until delivery
  Percentage of participants who intend to use similar method in future
Feeling alone during induction | At the time of recruitment until delivery
  Percentage of participants who felt lonely during induction
Duration of sleep | At the time of recruitment until delivery
  Duration of sleep during induction in hours
Able to rest and relax | At the time of recruitment until delivery
  Percentage of participants who are able to rest and relax
Feeling of unsafe during cervical ripening | At the time of recruitment until active phase of labour
  Percentage of participants who felt unsafe during cervical ripening
Embarrassed by the method | At the time of recruitment until active phase of labour
  Percentage of participants who felt embarrassed by the method

CONTACTS AND LOCATIONS:
Locations (1):
- UKM Medical Centre, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No